CLINICAL TRIAL: NCT07294300
Title: A Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of QLS2313 for Injection in Patients With Relapsed/Refractory Hematological Malignancies
Brief Title: A Phase I Trial of QLS2313 Injection in Relapsed/Refractory Hematological Malignancies
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QLS2313-101
Record Dates: First submitted 2025-12-08; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Relapsed/Refractory Hematological Malignancies
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- QLS2313 (Experimental)
  Interventions: Drug: QLS2313

INTERVENTIONS:
Drug: QLS2313 — CD79b/CD3/CD20;first in human; subcutaneous injection

SUMMARY:
This study is an open-label, dose-escalation and efficacy-expansion Phase I clinical trial to evaluate the safety, tolerability, PK profile, immunogenicity, and preliminary antitumor activity of QLS2313 as a monotherapy in patients with relapsed/refractory hematological malignancies.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females aged ≥ 18 years；
2. Patients with relapsed/refractory hematological malignancies, specifically patients with B-cell NHL or CLL/small lymphocytic lymphoma (SLL) as defined by the 2022 World Health Organization (WHO) classification, who are relapsed/refractory and have no standard of care available as judged by the investigator;
3. Having a measurable disease defined by appropriate disease response criteria;
4. Subjects with sufficient organ function prior to the first dose of the investigational drug
5. Eastern Cooperative Oncology Group (ECOG) performance status (PS) score: 0 or 1

Exclusion Criteria:

1. Previous treatment with a CD79b/CD3/CD20 trispecific antibody；
2. Known central nervous system (CNS) involvement；
3. Known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation/bone marrow transplantation；
4. Treatment with autologous stem cell transplantation within 3 months;
5. Prior genetically modified adoptive cell therapy (e.g., chimeric antigen receptor T cells [CAR-T] and natural killer cells [CAR-NK]) within 3 months
6. Presence of viral, bacterial or uncontrolled fungal infection requiring intravenous drug infusion within 1 week prior to the first dose
7. Presence of chronic or acute active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection, defined as HBV-5 test at screening indicating active infection (positive HBsAg and/or positive HBcAb) with HBV-DNA > ULN, or positive HCVAb and positive HCV-RNA, allowed for antiviral therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
DLT, MTD, RPIbD, and RP2D | to 2 years
  To evaluate the tolerability and safety of subcutaneously administered QLS2313 for Injection in patients with hematological malignancies, and to determine the MTD, RPIbD, and RP2D.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Jiaotong University School of Medicine Ruijin Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided